CLINICAL TRIAL: NCT03290417
Title: Correlative Analysis of the Genomics of Vitamin D and Omega-3 Fatty Acid Intake in Men Managed With Active Surveillance for Prostate Cancer
Brief Title: Correlative Analysis of the Genomics of Vitamin D and Omega-3 Fatty Acid Intake in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3816
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: Active Surveillance; Vitamin D; Omega-3 Fatty Acid; tumeric curcumin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin D; Cholecalciferol; Docosahexaenoic Acids; Curcumin

STUDY DESIGN:
Intervention Model Description: Parallel groups, one with a control diet, the other with a modified diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unmodified Diet (No Intervention): Patients are under active surveillance with no modification to their diet, as is standard of care for low risk prostate cancer
- Diet modification (Experimental): Patients receive Vitamin D, Omega-3 and turmeric curcumin as dietary supplements
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Omega-3; Dietary Supplement: Turmeric

INTERVENTIONS:
Dietary Supplement: Vitamin D — 5000 IU/cap; One cap by mouth daily
  Other Names: Vitamin D3
  Arms: Diet modification
Dietary Supplement: Omega-3 — 720 mg/cap; one capsule by mouth 3 times per day
  Other Names: Omegagenics
  Arms: Diet modification
Dietary Supplement: Turmeric — 250mg/cap; two capsules by mouth 4 times per day
  Other Names: Turmeric curcumin
  Arms: Diet modification

SUMMARY:
The purpose of this study is to see if eating vitamin D, omega 3 and turmeric (curcumin) slows the growth of prostate cancer in men on active surveillance.

DETAILED DESCRIPTION:
The primary objective is to investigate the influence of vitamin D, omega-3 fatty acids, and turmeric curcumin intake on the genomic landscape of NCCN very low and low risk patients managed with Active Surveillance. This will be measured by using genomic signatures in Decipher GRID and using the mixed effect linear model that tests for the interaction of treatment arm and time (base-line, 6 month and 12 month time points) with gene expression as the response variable.

The secondary objective is to evaluate prostate cancer aggressiveness pre and post intervention by looking at genes and gene signatures associated with vitamin D and omega-3 fatty acids pathways. Prognostic performance of GRID gene signatures will be evaluated using Active Surveillance 'Failure' (deferred treatment) as an additional endpoint.

The exploratory objective is to be able to use predictive genes and/or genomic signatures to assess benefit from vitamin D, omega-3 fatty acid and turmeric curcumin intake. This will only be possible once sufficient patient follow up is available.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the diagnosis of prostate cancer and be on active surveillance. For the purpose of this study, Active surveillance implies prostate-specific antigen (PSA)<10 ng/mL, biopsy Gleason sum </=6 with no pattern 4 or 5, cancer involvement of <33% of biopsy cores, and clinical stage T1/T2a tumor.
* Subjects must be followed at the Cleveland Clinic for active surveillance.
* Subjects must be willing to adhere to the dietary modification outlined in the protocol.
* Subjects must be willing to have prostate biopsies at the baseline, and six months after enrollment into the protocol
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects receiving any treatment other than AS for prostate cancer.
* Subjects not followed by the Cleveland Clinic.
* Subjects unable to adhere to the dietary modification outlined in the protocol.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
gene expression of very low and low risk prostate cancer patients on Active Surveillance | Up to 6 months
  The primary objective is to investigate the influence of vitamin D, omega-3 fatty acids, and turmeric curcumin intake on the genomic landscape of NCCN very low and low risk patients managed with Active Surveillance. This will be measured by using genomic signatures in Decipher GRID and using the mixed effect linear model that tests for the interaction of treatment arm and time
gene expression of very low and low risk prostate cancer patients on Active Surveillance | Up to 12 months
  The primary objective is to investigate the influence of vitamin D, omega-3 fatty acids, and turmeric curcumin intake on the genomic landscape of NCCN very low and low risk patients managed with Active Surveillance. This will be measured by using genomic signatures in Decipher GRID and using the mixed effect linear model that tests for the interaction of treatment arm and time

SECONDARY OUTCOMES:
Active Surveillance Failure | Up to 12 months
  Cox proportional hazards model will be used to study if genes are significantly predictive of this outcome. P-values will be corrected for multiple testing using the Benjamini-Hochberg procedure. Genes will be considered significant if the corresponding p-value is below 0.05 using a two-sided test.
Time to Active Surveillance Failure | Up to 12 months
  Time to event will be defined as time from enrollment into the study. P-values will be corrected for multiple testing using the Benjamini-Hochberg procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David Levy, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States